CLINICAL TRIAL: NCT02671500
Title: A Phase 3, Multicenter, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir/GS-5816 Fixed Dose Combination for 12 Weeks in Subjects With Chronic HCV
Brief Title: Efficacy and Safety of Sofosbuvir/Velpatasvir Fixed Dose Combination for 12 Weeks in Participants With Chronic HCV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-1518
Record Dates: First submitted 2016-01-29; First posted 2016-02-02 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SOF/VEL (Experimental): SOF/VEL FDC for 12 weeks
  Interventions: Drug: SOF/VEL

INTERVENTIONS:
Drug: SOF/VEL — SOF/VEL (400/100 mg) FDC tablet administered orally once daily
  Other Names: GS-7977/GS-5816; Epclusa®

SUMMARY:
The primary objectives of this study are to evaluate the efficacy, safety, and tolerability of treatment with sofosbuvir (SOF)/velpatasvir (VEL; GS-5816) fixed-dose combination (FDC) for 12 weeks in participants with chronic hepatitis C virus (HCV) infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent
* HCV RNA ≥ 10^4 IU/mL at screening
* Chronic HCV infection (≥ 6 months) documented by prior medical history or liver biopsy
* Any HCV genotype (1, 2, 3, 4, 5, 6 or indeterminate)
* HCV treatment-naive or treatment-experienced
* Liver imaging within 6 months of Day 1 is required in cirrhotic patients only to exclude hepatocellular carcinoma (HCC)

Key Exclusion Criteria:

* Current or prior history of clinically-significant illness (other than HCV), gastrointestinal disorder, clinical hepatic decompensation, or post-operative condition that could interfere with the absorption of the study drug
* Pregnant or nursing female or male with pregnant female partner
* Chronic liver disease of a non HCV etiology
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2016-04-19 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (38):
- China (25):
  - Beijing Ditan Hospital, Chaoyang, Beijing Municipality
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Tongji Hospital Affiliated to Tongji Medicine University, Wuhan, Hubei
  - Xiangyan Hospital, Central South University, Changsha, Hunan
  - Shanghai Public Health Clinical Center, Hongkou, Shanghai Municipality
  - Shanghai Ruijin Hospital, Huangpu, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Friendship Hospital Affiliate of Capital Medical University, Beijing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Guangzhou Eighth People's Hospital, Guangdong
  - The People's Hospital of Hainan Province, Hainan
  - The 2nd Xiangya Hospital of Central South University, Hunan
  - The Second Hospital of Nanjing, Jiangsu
  - The First Hospital of Jilin University, Jilin
  - Jinan Infectious Disease Hospital, Jinan
  - Shengjing Hospital of China Medical University, Liaoning
  - The First Affiliated Hospital of NanChang University, Nanchang
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Renji Hospital, Shanghai
  - The 3rd Hospital of Hebei Medical University, Shijiazhuang
  - Henan Province People's Hospital, Zhengzhou
- Malaysia (2):
  - University of Malaya, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuala Pahang
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
- Thailand (5):
  - Chulalongkorn Hospital, Bangkok
  - Ramathibodi Hospital Mahidol University, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakhon Chiangmai Hospital, Chiang Mai
  - Songklanagarind Hospital, Songkhla
- Vietnam (4):
  - Bach Mai Hospital, Hanoi
  - National Hospital for Tropical Disease, Hanoi
  - Ho Chi Minh City Hospital for Tropical Diseasees, Ho Chi Minh City
  - People's Hospital 115, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Lim SG, Rosmawati M, Phuong L, Hoi PT, McNabb BL, Lu S, et al. Safety and Efficacy of Sofosbuvir/Velpatasvir in a Genotype 1-6 HCV Infected Population from Singapore, Malaysia, Thailand, and Vietnam: Results from a Phase 3, Clinical Trial [Abstract 1094]. Hepatology 2017; 66 (1 Suppl): 586A.
- [Result] Wei L, Xie Q, Huang Y, Wu S, Xu M, Tang H, et al. Safety and Efficacy of Sofosbuvir/Velpatasvir in Genotype 1-6 HCV-Infected Patients in China: Results from a Phase 3 Clinical Trial. [Abstract 637]. Hepatology 2018; 68 (1 Suppl): 379A.
- [Derived] Wei L, Lim SG, Xie Q, Van KN, Piratvisuth T, Huang Y, Wu S, Xu M, Tang H, Cheng J, Le Manh H, Gao Y, Mou Z, Sobhonslidsuk A, Dou X, Thongsawat S, Nan Y, Tan CK, Ning Q, Tee HP, Mao Y, Stamm LM, Lu S, Dvory-Sobol H, Mo H, Brainard DM, Yang YF, Dao L, Wang GQ, Tanwandee T, Hu P, Tangkijvanich P, Zhang L, Gao ZL, Lin F, Le TTP, Shang J, Gong G, Li J, Su M, Duan Z, Mohamed R, Hou JL, Jia J. Sofosbuvir-velpatasvir for treatment of chronic hepatitis C virus infection in Asia: a single-arm, open-label, phase 3 trial. Lancet Gastroenterol Hepatol. 2019 Feb;4(2):127-134. doi: 10.1016/S2468-1253(18)30343-1. Epub 2018 Dec 14. PMID 30555048

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Asia. The first participant was screened on 19 April 2016. The last study visit occurred on 27 March 2018.
Pre-assignment Details: 437 participants were screened.
Groups:
- SOF/VEL: Sofosbuvir/velpatasvir (SOF/VEL) (400/100 mg) fixed-dose combination (FDC) tablet orally once daily for 12 weeks
Period: Overall Study
Arm/Group | SOF/VEL
Started | 375
Completed | 361
Not Completed | 14
Not completed — Lack of Efficacy | 12
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who were enrolled into the study and received at least 1 dose of study drug.
Groups:
- SOF/VEL: SOF/VEL (400/100 mg) FDC tablet orally once daily for 12 weeks.
Arm/Group | SOF/VEL
Number analyzed (Participants) | 375
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178
  Male | 197
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 374
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 375
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Vietnam | 36
  Singapore | 22
  China | 264
  Malaysia | 12
  Thailand | 41
HCV genotype [Count of Participants; unit: Participants]
  Genotype 1 | 129
  Genotype 2 | 64
  Genotype 3 | 84
  Genotype 6 | 98
IL28b Status [Count of Participants; unit: Participants]
  CC | 320
  CT | 53
  TT | 2
HCV RNA (log10 international units per milliliter [IU/mL]) [Mean (Standard Deviation); unit: log10 IU/mL] | 6.2 (0.86)
HCV RNA Category [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    < 800,000 IU/mL | 116
    ≥ 800,000 IU/mL | 259

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set included participants who were enrolled into the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SOF/VEL (Overall): All participants received SOF/VEL (400/100 mg) FDC tablet orally once daily for 12 weeks.
- SOF/VEL (China - Region 1): All participants in China received SOF/VEL (400/100 mg) FDC tablet orally once daily for 12 weeks.
- SOF/VEL (Southeast Asia - Region 2): All participants in Southeast Asia (Malaysia, Singapore, Thailand, and Vietnam) received SOF/VEL (400/100 mg) FDC tablet orally once daily for 12 weeks.
Arm/Group | SOF/VEL (Overall) | SOF/VEL (China - Region 1) | SOF/VEL (Southeast Asia - Region 2)
Number analyzed (Participants) | 375 | 264 | 111
Percentage of participants | 96.5 [94.1 to 98.1] | 96.2 [93.1 to 98.2] | 97.3 [92.3 to 99.4]
Statistical Analysis 1: Comparison: SOF/VEL (China - Region 1); A sample size of 260 participants in Region 1 would provide more than 80% power to detect an improvement of at least 6 percentage points in SVR12 rate from the performance goal of 85% by using a two-sided exact one-sample binomial test at the significance level of 0.05; Test type: Superiority; p < 0.001, 2-sided 1 sample exact binomial test

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Groups:
- SOF/VEL: SOF/VEL (400/100 mg) fixed-dose combination (FDC) tablet orally once daily for 12 weeks
Arm/Group | SOF/VEL
Number analyzed (Participants) | 375
Percentage of participants | 0

3. Secondary Outcome: Percentage of Participants With SVR at 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 375
Percentage of participants | 97.1 [94.8 to 98.5]

4. Secondary Outcome: Percentage of Participants With SVR at 24 Weeks After Discontinuation of Therapy (SVR24)
Description: SVR 24 was defined as HCV RNA < LLOQ at 24 weeks after stopping study treatment.
Time Frame: Posttreatment Week 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 375
percentage of participants | 96.5 [94.1 to 98.1]

5. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ On Treatment
Time Frame: Weeks 1, 2, 4, 6, 8, 10, and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 375
Percentage of participants
  Week 1 | 27.7 [23.3 to 32.6]
  Week 2: number analyzed (Participants) | 374
  Week 2 | 73.8 [69.0 to 78.2]
  Week 4: number analyzed (Participants) | 374
  Week 4 | 95.5 [92.8 to 97.3]
  Week 6: number analyzed (Participants) | 374
  Week 6 | 99.7 [98.5 to 100.0]
  Week 8: number analyzed (Participants) | 374
  Week 8 | 100.0 [99.0 to 100.0]
  Week 10: number analyzed (Participants) | 374
  Week 10 | 100.0 [99.0 to 100.0]
  Week 12: number analyzed (Participants) | 374
  Week 12 | 100.0 [99.0 to 100.0]

6. Secondary Outcome: Change From Baseline in HCV RNA
Time Frame: Baseline and up to Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL
Number analyzed (Participants) | 374
log10 IU/mL
  Change at Week 1: number analyzed (Participants) | 369
  Change at Week 1 | -4.38 (0.705)
  Change at Week 2: number analyzed (Participants) | 371
  Change at Week 2 | -4.89 (0.822)
  Change at Week 4 | -5.02 (0.849)
  Change at Week 6 | -5.03 (0.857)
  Change at Week 8 | -5.03 (0.857)
  Change at Week 10 | -5.03 (0.857)
  Change at Week 12 | -5.03 (0.857)

7. Secondary Outcome: Percentage of Participants With Overall Virologic Failure
Description: Virologic failure was defined as: (1) On-treatment virologic failure: Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment) or (2) Virologic relapse: confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL
Number analyzed (Participants) | 375
percentage of participants | 3.2

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set included participants who were enrolled into the study and received at least 1 dose of study drug.
Groups:
- SOL/VEL: SOL/VEL (400/100 mg) FDC tablet orally once daily for 12 weeks.
Arm/Group | SOL/VEL
All-Cause Mortality (participants affected / at risk) | 0/375
Serious Adverse Events (participants affected / at risk) | 3/375
Other Adverse Events (participants affected / at risk) | 36/375
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOL/VEL (N=375)
Diabetic foot infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOL/VEL (N=375)
Upper respiratory tract infection (Infections and infestations) | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol: Original (2015-01-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT02671500/Prot_000.pdf
  • Study Protocol: Amendment 1 (2015-04-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT02671500/Prot_001.pdf
  • Statistical Analysis Plan (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT02671500/SAP_002.pdf